CLINICAL TRIAL: NCT00443027
Title: Effect Of Menstrual Cycle On Vaginal Blood Flow (As Determined By The Heat Wash-Out Technique) Before, During And After Visual Sexual Stimulation In Pre-Menopausal Healthy Women.
Brief Title: Effect Of Menstrual Cycle On Vaginal Blood Flow In Pre-Menopausal Healthy Women.
Acronym: HWO VBF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A9001303
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Sexual Dysfunction, Physiological
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaginal Heat Wash-Out Device (Experimental)
  Interventions: Device: Vaginal Heat Wash-Out Device

INTERVENTIONS:
Device: Vaginal Heat Wash-Out Device — No drug administered. Device tested three times with each subject.

SUMMARY:
The Pfizer developed Heat Wash-Out (HWO) system is a software controlled electromechanical system designed to measure vaginal wall blood flow. A small vaginal probe is attached to a control unit. Output data is collected on a PC. By measuring the clearance of heat from the heated probe, a direct measure of absolute blood flow can be obtained. The study will assess changes in vaginal blood flow across the menstrual cycle following visual sexual stimulation.

DETAILED DESCRIPTION:
Medical Device Development

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal healthy women aged 18-45 with regular, natural menstrual cycles.
* Subjects must be void of Female Sexual Disorder.

Exclusion Criteria:

* Pregnant or lactating women
* Postmenopausal subjects
* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric or neurologic disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To investigate differences in vaginal blood flow across the menstrual cycle following visual sexual stimulation. | 28d
To assess the safety and toleration of the heat washout device. | 28d

SECONDARY OUTCOMES:
To investigate changes in subjective acute sexual arousal following visual sexual stimulation across the menstrual cycle. | 28d

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Australia (2):
  - Pfizer Investigational Site, Dulwich, South Australia
  - Pfizer Investigational Site, Nedlands, Western Australia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001303&StudyName=Effect%20Of%20Menstrual%20Cycle%20On%20Vaginal%20Blood%20Flow%20In%20Pre-Menopausal%20Healthy%20Women.